CLINICAL TRIAL: NCT03337529
Title: Restless Legs Syndrome in Hemodialysis Patients: Prevalence, Associated Risk Factors and Efficacy of Vitamin C as a Treatment
Brief Title: Restless Legs Syndrome in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Hania Jarkas, neurologist, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 10082017
Record Dates: First submitted 2017-11-06; First posted 2017-11-09 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Restless Leg Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin C (Experimental): RLS positive patients will be assessed for the severity. They will be given 200 mg Vitamin C for 8 weeks duration. Patients will be re-assessed for the severity of restless leg syndrome.
  Interventions: Other: Vitamin C
- Placebo (Placebo Comparator): RLS positive patients will be assessed for the severity. They will be given 200 mg placebo for 8 weeks duration. Patients will be re-assessed for the severity of restless leg syndrome.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Vitamin C — 200 mg Vitamin C will be given on daily basis for 8 weeks
  Arms: Vitamin C
Other: Placebo — 200 mg placebo will be given on daily basis for 8 weeks
  Arms: Placebo

SUMMARY:
Restless legs syndrome (RLS) is defined as the spontaneous movement of the limbs (mainly legs) associated with unpleasant - painful sensation which is relieved by moving the affected limb. It is a common disorder in hemodialysis patients that leads to insomnia, impaired daytime functioning and quality of life. Symptoms of RLS are estimated to affect up to 25% of patients on dialysis when the international RLS diagnostic criteria are applied. Various pharmacological and non-pharmacological interventions have been used to treat primary RLS. However, the evidence for use of these interventions in people with End stage renal disease is not well established; and some have serious side effects. Because high oxidative stress has been implicated in the pathogenesis of RLS, investigators thought of evaluating the efficacy of vitamin C in reducing the severity of RLS symptoms in hemodialysis patients in this randomized, double-blind, placebo-controlled, two arm parallel trial. To note that only two studies were done worldwide that proved the efficacy of vitamin C in those patients.

DETAILED DESCRIPTION:
The investigators are proposing to carry out a clinical trial. Around 100 stable hemodialysis adult patients at Makassed general hospital dialysis center and around 150 patients at Sahel general hospital and Zahraa hospital will be assessed according to the international RLS criteria. The data on individual, clinical and laboratory indices will be obtained from patients' recorded files and interviews. The investigators will compare the RLS group versus the non RLS group according to these factors to find the independently associated factors for RLS in dialysis patients.

Those who fulfill all four diagnostic criteria for RLS (confirmed independently by 2 neurologists) will be classified as "RLS positive" and will be asked to answer 10 questions on the international RLS study group (IRLSSG) rating scale. The IRLSSG rating scale was also used to evaluate the severity of RLS symptoms. These patients will be randomly allocated to two parallel groups to receive vitamin C (200 mg) or placebo for eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* patients under regular hemodialysis
* with no acute illness
* not hospitalized

Exclusion Criteria:

* Patients receiving:
* tricyclic antidepressants,
* selective serotonin reuptake inhibitors,
* dopamine antagonists,
* dopamine blocking,
* antiemetics,
* lithium,
* sedative antihistamines,
* Patients with a history of renal stones

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2018-04-15 (Actual)

PRIMARY OUTCOMES:
change in the international restless legs syndrome (IRLS) rating scale score | 8 weeks
  change in the IRLS rating scale sum score from baseline to the end of treatment.The scale ranges between 0 and 40 which is the total score. A score between 31 and 40, indicates very severe RLS. A score between 21 and 30 indicates severe RLS. A score between 11 and 20 indicates moderate RLS. A score between 1 and 10 indicates mild RLS and a score of 0 means no RLS.

SECONDARY OUTCOMES:
incidence of RLS | 8 weeks
  identify the incidence of restless legs syndrome in end stage renal disease (ESRD) patients on dialysis in Lebanon
Risk factors | 8 weeks
  identify risk factors associated with RLS

CONTACTS AND LOCATIONS:
Overall Officials: Hania Jarkas, MD, Principal Investigator — Makassed General Hospital
Locations (1):
- Makassed General Hospital, Beirut, Lebanon